CLINICAL TRIAL: NCT05995743
Title: Aerobic Physical Fitness and Health-related Quality of Life in Children With Sickle Cell Disease.
Brief Title: VO2max & HRQoL in Children With Sickle Cell Disease
Acronym: VO2drépano
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0192
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Sickle Cell; Children
Keywords: Cardiopulmonary exercise test; VO2max; Sickle cell disease; Child; Heath-related quality of life; Cardiopulmonary rehabilitation
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children with sickle cell disease: Children aged 6 to 17 years with a confirmed diagnosis of sickle cell disease (i.e., homozygous HbS/S or heterozygous HbS/C mutations)
- Controls: Healthy children referred for a non-severe functional symptom linked to exercise: Children aged 6 to 17 years with a completely normal check-up, including physical examination, ECG, echocardiography, and spirometry. Children with any chronic disease, medical condition, or medical treatment and those requiring any further specialized medical consultation were not eligible.

SUMMARY:
Sickle cell disease is the most common inherited genetic disorder, accounting for 300,000 births worldwide per year. It is caused by an autosomal recessive mutation of the β-globin gene, responsible for an abnormal hemoglobin, the main protein in red blood cells, responsible for transporting oxygen from the lungs to the tissues. The abnormal hemoglobin, known as "Sickle" or S, deforms the red blood cell, causing chronic hemolytic anemia, organ damage (heart, spleen, etc.) and vaso-occlusive crises. Therapeutic progress and specialised patient follow-up have considerably improved the vital and functional prognosis of children and adolescents with sickle cell disease. Physical fitness, measured during a cardiorespiratory exercise test (CPET), is used to determine maximal oxygen uptake (VO2max). Patients with sickle cell disease have a multifactorial limitation of exercise tolerance, which may affect their physical fitness. Authors have shown that VO2max is impaired in children and adolescents with sickle cell disease, independently of their baseline hemoglobin level. Yet VO2max is a key determinant of health-related quality of life (HRQoL) in patients being monitored for a chronic disease. In the past, our team has contributed to the assessment of HRQoL in several groups of pediatric patients suffering from chronic disease (congenital heart disease, PAH). To date, the link between impaired physical fitness and HRQoL has not been demonstrated in sickle cell children. The pathophysiological determinants of reduced physical capacity and exercise tolerance in sickle cell patients have also not been fully elucidated. Studying these factors will enable us to propose appropriate treatment in the future, with the aim of improving physical fitness and HRQoL in children and adolescents with sickle cell disease.

DETAILED DESCRIPTION:
This prospective case-control study included sickle cell children and healthy controls from 6 to 17 years old. Patients refuse the use of medical data will be excluded.

After description of the study sample, we will first compare the VO2max Z-score between cases and controls. We will correlate the VO2max to PedsQL self- and proxy-related and Ricci and Gagnon scores (use of the coefficient of correlation rhô). Then we will compare others CPET parameters and will determine associated factors of VO2max with others resting data : hematological, respiratory, cardiologic, anthropometric, educational (use of the coefficient of correlation rhô, and multivariate linear regression model).

ELIGIBILITY:
Sickle cell children

Inclusion Criteria:

* Child from 6 to 17 years old, with a confirmed diagnosis of sickle cell disease (i.e., homozygous HbS/S or heterozygous HbS/C mutations), during their routine follow-up, having performed :
* a hematology consultation : physical examination, blood test
* a cardiology consultation : electrocardiogram, transthoracic echocardiography
* a respiratory plethysmography
* a CPET and to fill in the study questionnaires.

Exclusion Criteria:

* Parents' refusal to use medical data.

Healthy children

Inclusion Criteria:

* Child from 6 to 17 years old having performed a cardio-respiratory exercise test for chest pain, dyspnea on exertion, heart murmur and whose results do not find:
* Congenital heart disease (normal echocardiography and ECG)
* Respiratory disease (normal FEV1 and FVC)
* Child having performed a maximal cardio-respiratory stress exercise until exhaustion.

Exclusion Criteria:

* Child taking long-term drug treatment
* Child with chronic disease
* Parents' refusal to use medical data.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sickle cell children cohort consisted of children with a genetic diagnosis of sickle cell disease (HbS/S or HbS/C), followed at the Department of Pediatrics of Montpellier University Hospital, a tertiary care academic institution in southern France.
  Healthy children cohort consisted of children referred to a pediatric cardiologist for a nonsevere functional symptom related to exercise (murmur, palpitation, chest pain, and dyspnoea) or for a medical sports certificate. These children needed to have a completely normal check-up, including physical examination, ECG, and echocardiography. Children with any chronic disease, medical condition or medical treatment, and those requiring any further specialized medical consultation were not eligible.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Difference between aerobic fitness evaluated by VO2max, expressed in Z-score between cases and controls | 1 day

SECONDARY OUTCOMES:
Correlation between aerobic fitness and quality of life in cases group | 1 day
  To analyze this, we will correlate the VO2max Z-score and the assessment of health-related quality of life (measured by PedQL 4.0).
Correlation between aerobic fitness and physical activity level, in cases group | 1 day
  To analyze this, we will correlate the VO2max Z-score and the assessment of physical activity level (measured by Ricci and Gagnon questionnaire).
Correlation between aerobic fitness and educational level (knowledge about disease), in cases group | 1 day
  To analyze this, we will correlate the VO2max Z-score and the assessment of educational level (local disease knowledge questionnaire).
Correlation between aerobic fitness and VO2max limiting factors in cases group: demographic, genetic mutation, clinical (comorbidities, respiratory function, cardiac function, anemia, CPET data) | 1 day
  To analyze this, we will correlate the VO2max Z-score and demographic data, genetic mutation, spirometry, plethysmography, trans-thoracic echocardiography, hemoglobin level, other CPET data.

CONTACTS AND LOCATIONS:
Overall Officials: Corentin Laurent-Lacroix, Resident, Principal Investigator — Montpellier University Hospital
Locations (1):
- Pediatric and Congenital Cardiology Department, Arnaud De Villeneuve University Hospital, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piel FB, Steinberg MH, Rees DC. Sickle Cell Disease. N Engl J Med. 2017 Apr 20;376(16):1561-1573. doi: 10.1056/NEJMra1510865. No abstract available. PMID 28423290
- [Background] Ferraresi M, Panzieri DL, Leoni S, Cappellini MD, Kattamis A, Motta I. Therapeutic perspective for children and young adults living with thalassemia and sickle cell disease. Eur J Pediatr. 2023 Jun;182(6):2509-2519. doi: 10.1007/s00431-023-04900-w. Epub 2023 Mar 31. PMID 36997768
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- [Background] Connes P, Machado R, Hue O, Reid H. Exercise limitation, exercise testing and exercise recommendations in sickle cell anemia. Clin Hemorheol Microcirc. 2011;49(1-4):151-63. doi: 10.3233/CH-2011-1465. PMID 22214686
- [Background] Panepinto JA, O'Mahar KM, DeBaun MR, Loberiza FR, Scott JP. Health-related quality of life in children with sickle cell disease: child and parent perception. Br J Haematol. 2005 Aug;130(3):437-44. doi: 10.1111/j.1365-2141.2005.05622.x. PMID 16042695
- [Background] Liem RI, Reddy M, Pelligra SA, Savant AP, Fernhall B, Rodeghier M, Thompson AA. Reduced fitness and abnormal cardiopulmonary responses to maximal exercise testing in children and young adults with sickle cell anemia. Physiol Rep. 2015 Apr;3(4):e12338. doi: 10.14814/phy2.12338. PMID 25847915
- [Background] Callahan LA, Woods KF, Mensah GA, Ramsey LT, Barbeau P, Gutin B. Cardiopulmonary responses to exercise in women with sickle cell anemia. Am J Respir Crit Care Med. 2002 May 1;165(9):1309-16. doi: 10.1164/rccm.2002036. PMID 11991885
- [Background] Woodson RD. Hemoglobin concentration and exercise capacity. Am Rev Respir Dis. 1984 Feb;129(2 Pt 2):S72-5. doi: 10.1164/arrd.1984.129.2P2.S72. No abstract available. PMID 6696347
- [Background] Pianosi P, D'Souza SJ, Esseltine DW, Charge TD, Coates AL. Ventilation and gas exchange during exercise in sickle cell anemia. Am Rev Respir Dis. 1991 Feb;143(2):226-30. doi: 10.1164/ajrccm/143.2.226. PMID 1990932
- [Background] Klings ES, Wyszynski DF, Nolan VG, Steinberg MH. Abnormal pulmonary function in adults with sickle cell anemia. Am J Respir Crit Care Med. 2006 Jun 1;173(11):1264-9. doi: 10.1164/rccm.200601-125OC. Epub 2006 Mar 23. PMID 16556694
- [Background] Olorunyomi OO, Liem RI, Hsu LL. Motivators and Barriers to Physical Activity among Youth with Sickle Cell Disease: Brief Review. Children (Basel). 2022 Apr 17;9(4):572. doi: 10.3390/children9040572. PMID 35455616
- [Background] Amedro P, Gavotto A, Guillaumont S, Bertet H, Vincenti M, De La Villeon G, Bredy C, Acar P, Ovaert C, Picot MC, Matecki S. Cardiopulmonary fitness in children with congenital heart diseases versus healthy children. Heart. 2018 Jun;104(12):1026-1036. doi: 10.1136/heartjnl-2017-312339. Epub 2017 Nov 23. PMID 29170358
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Abassi H, Gavotto A, Picot MC, Bertet H, Matecki S, Guillaumont S, Moniotte S, Auquier P, Moreau J, Amedro P. Impaired pulmonary function and its association with clinical outcomes, exercise capacity and quality of life in children with congenital heart disease. Int J Cardiol. 2019 Jun 15;285:86-92. doi: 10.1016/j.ijcard.2019.02.069. Epub 2019 Mar 1. PMID 30857849
- [Background] Amedro P, Basquin A, Gressin V, Clerson P, Jais X, Thambo JB, Guerin P, Cohen S, Bonnet D. Health-related quality of life of patients with pulmonary arterial hypertension associated with CHD: the multicentre cross-sectional ACHILLE study. Cardiol Young. 2016 Oct;26(7):1250-9. doi: 10.1017/S1047951116000056. Epub 2016 Mar 16. PMID 26980152
- [Background] Das BB, Sobczyk W, Bertolone S, Raj A. Cardiopulmonary stress testing in children with sickle cell disease who are on long-term erythrocytapheresis. J Pediatr Hematol Oncol. 2008 May;30(5):373-7. doi: 10.1097/MPH.0b013e318165b298. PMID 18458572
- [Background] Gavotto A, Mura T, Rhodes J, Yin SM, Hager A, Hock J, Guillaumont S, Vincenti M, De La Villeon G, Requirand A, Picot MC, Huguet H, Souilla L, Moreau J, Matecki S, Amedro P. Reference values of aerobic fitness in the contemporary paediatric population. Eur J Prev Cardiol. 2023 Jul 12;30(9):820-829. doi: 10.1093/eurjpc/zwad054. PMID 36809338
- [Background] Takken T, Blank AC, Hulzebos EH, van Brussel M, Groen WG, Helders PJ. Cardiopulmonary exercise testing in congenital heart disease: equipment and test protocols. Neth Heart J. 2009 Sep;17(9):339-44. doi: 10.1007/BF03086280. PMID 19949476
- [Background] Varni JW, Burwinkle TM, Seid M, Skarr D. The PedsQL 4.0 as a pediatric population health measure: feasibility, reliability, and validity. Ambul Pediatr. 2003 Nov-Dec;3(6):329-41. doi: 10.1367/1539-4409(2003)0032.0.co;2. PMID 14616041
- [Background] Amedro P, Huguet H, Macioce V, Dorka R, Auer A, Guillaumont S, Auquier P, Abassi H, Picot MC. Psychometric validation of the French self and proxy versions of the PedsQL 4.0 generic health-related quality of life questionnaire for 8-12 year-old children. Health Qual Life Outcomes. 2021 Mar 4;19(1):75. doi: 10.1186/s12955-021-01714-y. PMID 33663527
- [Background] Vuillemin A, Denis G, Guillemin F, Jeandel C. [A review of evaluation questionnaires for physical activity]. Rev Epidemiol Sante Publique. 1998 Feb;46(1):49-55. French. PMID 9533234
- [Background] Pianosi P, D'Souza SJ, Charge TD, Beland MJ, Esseltine DW, Coates AL. Cardiac output and oxygen delivery during exercise in sickle cell anemia. Am Rev Respir Dis. 1991 Feb;143(2):231-5. doi: 10.1164/ajrccm/143.2.231. PMID 1990933
- [Background] Powell AW, Alsaied T, Niss O, Fleck RJ, Malik P, Quinn CT, Mays WA, Taylor MD, Chin C. Abnormal submaximal cardiopulmonary exercise parameters predict impaired peak exercise performance in sickle cell anemia patients. Pediatr Blood Cancer. 2019 Jun;66(6):e27703. doi: 10.1002/pbc.27703. Epub 2019 Mar 7. PMID 30848046
- [Background] Amedro P, Gavotto A, Legendre A, Lavastre K, Bredy C, De La Villeon G, Matecki S, Vandenberghe D, Ladeveze M, Bajolle F, Bosser G, Bouvaist H, Brosset P, Cohen L, Cohen S, Corone S, Dauphin C, Dulac Y, Hascoet S, Iriart X, Ladouceur M, Mace L, Neagu OA, Ovaert C, Picot MC, Poirette L, Sidney F, Soullier C, Thambo JB, Combes N, Bonnet D, Guillaumont S. Impact of a centre and home-based cardiac rehabilitation program on the quality of life of teenagers and young adults with congenital heart disease: The QUALI-REHAB study rationale, design and methods. Int J Cardiol. 2019 May 15;283:112-118. doi: 10.1016/j.ijcard.2018.12.050. Epub 2018 Dec 20. PMID 30616811
- [Derived] Laurent-Lacroix C, Vincenti M, Matecki S, Mahe P, Moulis L, De La Villeon G, Guillaumont S, Requirand A, Moreau J, Lalande M, Picot MC, Amedro P, Gavotto A. Aerobic physical capacity and health-related quality of life in children with sickle cell disease. Pediatr Res. 2024 Sep;96(4):1006-1012. doi: 10.1038/s41390-024-03143-1. Epub 2024 Mar 15. PMID 38491141